CLINICAL TRIAL: NCT01742312
Title: Effect of Neoadjuvant Chemotherapy on Muscle Mass and Peri-operative Cardiorespiratory Performance in Patients Undergoing Oesophageal Cancer- a Pilot Study
Brief Title: Effects of Chemotherapy on Muscle Mass and Exercise Performance in Patients With Oesophageal Cancer.
Acronym: Oeso-Chemo
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 10/H0405/38
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Oesophageal Adenocarcinoma
Keywords: neoadjuvant chemotherapy; oesophageal cancer; cardiorespiratory performance
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Neoplasms | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood tests for serum albumin and total protien levels.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- oesophageal adenocarcinoma: DEXA scan cardio-pulmonary exercise testing (CPEX) muscle biopsy
  Interventions: Radiation: DEXA scan; Procedure: Muscle biopsy; Other: cardio-pulmonary exercise testing (CPEX)

INTERVENTIONS:
Radiation: DEXA scan — all patients will undertake a full body DEXA scan before and after chemotherapy
Procedure: Muscle biopsy — All patients will have a muscle biopsy before and after chemotherapy
Other: cardio-pulmonary exercise testing (CPEX) — patients will undertake exercise in the form of an exercise bike whilst having their cardiac and ventilatory performance analysed. This will take place before and after neoadjuvant chemotherapy

SUMMARY:
Curative treatment for oesophageal cancer involves undertaking chemotherapy followed by an operation to remove the tumour. Chemotherapy has several effects upon the body, including effects upon the systems that control the creation and breakdown of muscle. We aim to review these effects by recording changes in the amount of exercise patients are able to undertake after chemotherapy and reviewing changes in muscle mass.

DETAILED DESCRIPTION:
We aim to review the effects of chemotherapy on skeletal muscle mass and cardio-respiratory performance in patients with oesophageal adenocarcinoma. All patients will be assessed by a Consultant Anaesthetist and a medical member of the Research team before commencing chemotherapy and after finishing their course. These assessments include a nutritional assessment, performance status assessments, blood assays, dual energy X-ray absorptiometry (DEXA) scans, cardio-pulmonary exercise (CPEX) testing and a muscle biopsy.

ELIGIBILITY:
Inclusion Criteria:

* oesophageal cancer
* Multidisciplinary team decision to offer neoadjuvant chemotherapy prior to surgery

Exclusion Criteria:

* Metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: healthy volunteers oesophageal cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
muscle mass | 3 months
  variations in muscle mass during neoadjuvant chemotherapy

SECONDARY OUTCOMES:
nutritional status | 3 months
  assess nutritional status post chemotherapy via serum protein levels.
all cause mortality | 3 months
  Evidence of mortality and relate this to aerobic ability.
mitochondrial function performance status | 3 months
  review changes in mitochondrial function after neoadjuvant chemotherapy
cardiorespiratory performance (peak VO2) | 3 months
  review changes in cardiorespiratory performance (peak VO2) after neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: John Williams, MBChB, FFPMRCA, PhD, Study Chair — Graduate Entry Medical School, University of Nottingham
Locations (1):
- Graduate Entry Medical School, University of Nottingham, Derby, Derbyshire, United Kingdom